CLINICAL TRIAL: NCT01873300
Title: Endoscopic Esophageal Myotomy for the Treatment of Achalasia
Brief Title: Endoscopic Myotomy for the Treatment of Achalasia (Motility Disorder) of the Esophagus - POEM Procedure
Acronym: POEM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David W. Rattner, MD, Professor of Surgery - Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011P001806
Record Dates: First submitted 2013-06-05; First posted 2013-06-10 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Achalasia
Keywords: Achalasia; Dysphagia; Endoscopic; Myotomy; Heller; NOTES; POEM
MeSH Terms: conditions — Esophageal Achalasia; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment group (Experimental): Patients undergoing POEM procedure
  Interventions: Procedure: Endoscopic Esophageal Myotomy

INTERVENTIONS:
Procedure: Endoscopic Esophageal Myotomy — Endoscopic mucosotomy, with submucosal tunneling and circular muscular fiber myotomy and mucosa closure.
  Other Names: POEM; Trans-esophageal endoscopic myotomy; Per-oral endoscopic myotomy; Endoscopic Heller Myotomy

SUMMARY:
Endoscopic Esophageal Myotomy (POEM), the research procedure, splits the lower esophageal sphincter muscle fibers from the inside of the esophagus, avoiding several abdominal incisions (belly area cuts), by using an endoscope to create a small cut at the most inner layer of the esophagus to expose the esophageal sphincter muscle fibers from the inside of the esophagus. The investigators are studying whether subjects who undergo Endoscopic Esophageal Myotomy will have similar functional outcome, and at the same time less pain, scar formation and wound infection than with laparoscopic or open surgery.

DETAILED DESCRIPTION:
The purpose of this research study is to find out more about a less invasive way of doing the surgical procedure (esophageal myotomy) to treat Achalasia.

Achalasia is a disease of the esophagus, where the lower esophageal sphincter fails to relax, causing difficulty in swallowing.

Esophageal myotomy (Heller myotomy) is surgically cutting the muscle fibers of the esophageal sphincter to allow passage of food into the stomach.

Esophageal myotomy is routinely done either by laparoscopic or open surgery. Laparoscopic surgery requires several (about 4 to 5) small incisions in the abdomen to allow the camera and surgical instruments to be introduced into the abdominal cavity to perform the myotomy. In open surgery, a 6- to 8-inch abdominal incision is made to gain access to the abdominal cavity to perform the myotomy.

Endoscopic Esophageal Myotomy (POEM), the research procedure, splits the lower esophageal sphincter muscle fibers from the inside of the esophagus, avoiding several abdominal incisions.

The researchers are investigating how safe Endoscopic Esophageal Myotomy is and how well it works. Additionally, the researchers will assess the level of pain and the amount of scarring subjects has after this surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of achalasia
* Age 18-65
* ASA class 1-2

Exclusion Criteria:

* Pregnant women
* Any prior surgical or endoscopic treatment for achalasia except dilation less than 20 mm
* Patients who are taking immunosuppressive medications or are immunocompromised Patients on blood thinners or aspirin or with history of bleeding disorders
* ASA class III patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Improvement of quality of life and dysphagia symptoms | 6 months
  Patients will be given a quality of life and dysphagia questionare before surgery and at 3 and 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: David W Rattner, MD, Principal Investigator — Massachusetts General Hospital; Ozanan R Meireles, MD, Study Director — Masschusetts General Hospital / Harvard Medical School
Locations (1):
- Masschusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Inoue H, Kudo SE. [Per-oral endoscopic myotomy (POEM) for 43 consecutive cases of esophageal achalasia]. Nihon Rinsho. 2010 Sep;68(9):1749-52. Japanese. PMID 20845759
- [Background] Inoue H, Tianle KM, Ikeda H, Hosoya T, Onimaru M, Yoshida A, Minami H, Kudo SE. Peroral endoscopic myotomy for esophageal achalasia: technique, indication, and outcomes. Thorac Surg Clin. 2011 Nov;21(4):519-25. doi: 10.1016/j.thorsurg.2011.08.005. PMID 22040634
- [Background] von Renteln D, Inoue H, Minami H, Werner YB, Pace A, Kersten JF, Much CC, Schachschal G, Mann O, Keller J, Fuchs KH, Rosch T. Peroral endoscopic myotomy for the treatment of achalasia: a prospective single center study. Am J Gastroenterol. 2012 Mar;107(3):411-7. doi: 10.1038/ajg.2011.388. Epub 2011 Nov 8. PMID 22068665